CLINICAL TRIAL: NCT01533337
Title: Free Dorsal Digital Flap for Reconstruction of Volar Soft Tissue Defect of Digits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tschen3886
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2024-01-22 (Actual); Status verified 2012-02

CONDITIONS: Nerve Injury; Digital Pulp Defect
Keywords: dorsal digital free flap; dorsal branch of proper digital nerve; dorsal branch of proper digital artery; proper digital artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- finger (Other): Free dorsal digital flap transferring is used for reconstruction of soft-tissue defects
  Interventions: Procedure: Free dorsal digital flap

INTERVENTIONS:
Procedure: Free dorsal digital flap — The dorsal digital flap, including both dorsal branches of the proper digital nerves, was designed on the dorsum of the donor finger between the distal third of the proximal phalanx and the distal interphalangeal joint.

SUMMARY:
The aim of the current report is to investigate the feasibility of transferring the free dorsal digital flap, including both dorsal branches of the proper digital nerves (PDNs), to reconstruct the volar soft tissue defect of digits. Sensory restoration of the reconstructed digit was evaluated via static two-point discrimination (2PD). The range of motion (ROM) of the donor middle and ring fingers was measured.

DETAILED DESCRIPTION:
Sensory restoration of the reconstructed digit was evaluated via static two-point discrimination (2PD). The range of motion (ROM) of the donor middle and ring fingers was measured. The data were compared with those of the contralateral, uninjured hand.

ELIGIBILITY:
Inclusion Criteria:

1. soft tissue defects in the fingertip, pulp, or volar surface of the digits;
2. a defect > 2 cm in length;
3. unavailability of the homodigital and heterodigital island flaps because of concomitant injuries to donor fingers; and
4. the patient refuses to use tissues from the toe.

Exclusion Criteria:

1. soft tissue defects in the dorsum of the digits;
2. a defect < 2 cm in length;
3. homodigital and heterodigital island flaps are available.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination (2PD) test | 25 months
  The test points were at the centers of the radial and ulnar portions of the digital pulp and the donor sites separately. Each area was tested 3 times with a Dellon-Mackinnon discriminator. Two out of 3 correct answers were considered proof of perception before proceeding to another lower value.